CLINICAL TRIAL: NCT01821313
Title: Effects of High Intensity Interval Exercise on Inflammation and Endothelial Function in Children & Adolescents With Obesity
Brief Title: CASH- Children Active to Stay Healthy
Acronym: CASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Ihuoma Eneli, Medical director/ Associate professor, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB12-00197
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Childhood Obesity; Inflammation
Keywords: Childhood obesity; Inflammation; Endothelial function; Exercise
MeSH Terms: conditions — Pediatric Obesity; Inflammation; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate exercise (Experimental): The subject will participate in a 6-week exercise intervention, 3 days per week on a cycle ergometer. The moderate exercise group will begin with a five-minute warm-up, cycling at 50-55% of the subject's maximal heart rate as determined by the initial fitness assessment. Following the warm-up, the moderate group will cycle for 30 minutes at 65-70% of maximal heart rate. The subject will then complete a 5-minute cool-down at 50-55% of maximal heart rate. Heart rate will be measured via individual heart rate monitors.
  Interventions: Other: Moderate exercise
- High Intensity Interval Exercise (HIIE) (Active Comparator): The subject will participate in a 6-week exercise intervention, 3 days per week on a cycle ergometer. The subjects in the HIIE group will begin with a five-minute warm-up at 50-55% of the subject's maximal heart rate as determined by the initial fitness assessment. Following the warm-up, the HIIE group will perform 10, two-minute exercise bouts at 90-95% of maximal heart rate, with one minute of active recovery at 55% of maximal heart rate between each interval for a total of 30 minutes. They will complete the test with a 5-minute cool-down at 50-55% of maximal heart rate. Heart rate will be measured via individual heart rate monitors.
  Interventions: Other: High Intensity Interval Exercise

INTERVENTIONS:
Other: Moderate exercise
  Arms: Moderate exercise
Other: High Intensity Interval Exercise
  Arms: High Intensity Interval Exercise (HIIE)

SUMMARY:
The purpose of this study is to examine the effects of high intensity interval exercise (HIIE) on inflammation and endothelial dysfunction found in children with obesity. Our working hypothesis is that, compared with obese children prescribed moderate exercise, obese children prescribed HIIE will demonstrate greater improvements in endothelial function and inflammatory markers following a 6-week exercise intervention.

DETAILED DESCRIPTION:
Obesity, even in children, is generally accompanied by a state of chronic inflammation. To combat childhood obesity, clinicians and scientists recommend lifestyle interventions that include increased physical activity and exercise in an attempt to promote weight loss and, consequently, decrease comorbidities associated with excess adiposity. More importantly, it appears that the influence of regular exercise may offer children with obesity a multitude of health benefits, independent of weight loss. However, the intensity of exercise required to elicit significant health benefits is still unclear. Therefore, the aim of the present project is to study the influence of high intensity interval exercise (HIIE) on the existing inflammatory state found in obesity. Specifically, the proposed project will examine endothelial function and markers of inflammation, such as TNFa, IL-6, hsCRP, and adiponectin, in children with obesity before and after an exercise intervention. The data will then be used to determine if changes in these values differ in magnitude based on the intensity of exercise. Children with obesity will be randomized into either moderate exercise or HIIE groups, and attend sessions 3 times per week for 6 weeks. The moderate group will cycle continuously for 30 minutes at 65%-70% of maximal heart rate and the HIIE group will perform ten, 2-minute bouts at 90%-95% of maximal heart rate. Outcome measures of body composition, aerobic capacity, blood lipids, glucose metabolism, endothelial function, and inflammation will be measured pre- and post-intervention. Results may help in establishing exercise protocols not only for children with obesity, but also other inflammatory diseases such as diabetes, cancer, and arthritis.

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years old
* obesity (defined as as BMI≥ 95th percentile for age and sex as defined by the Centers for Disease Control

Exclusion Criteria:

* active participation in ≥30 minutes of vigorous exercise more than 2 days per week
* participation in an organized combined diet/exercise weight loss intervention
* acute inflammatory disease or febrile illness
* recent trauma or injury
* asthma requiring steroid use or that has resulted in hospitalization within 3 months prior to enrollment
* chronic disease known to affect inflammation (e.g. lupus)
* any renal, heart, or liver disease

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Inflammation and endothelial function measured via forearm vascular resistance (FVR) and blood markers including tumor necrosis factor alpha (TNF-a), interleukin-6 (IL-6), adiponectin, high sensitivity C-reactive protein (hsCRP), and endothelin 1. | Within one month pre and one month post-intervention
  The primary outcomes are the percent change in FVR and in inflammatory markers (hsCRP, IL-6, TNF-α, and adiponectin) from pre- to post-intervention in both groups.

SECONDARY OUTCOMES:
Percent difference in inflammation and endothelial function between moderate and high intensity interval exercise (HIIE) groups. | Within one month pre- and no more than one month post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ihuoma Eneli, MD, Principal Investigator — Nationwide Children's Hospital; Andrea Bonny, MD, Principal Investigator — Nationwide Children's Hospital; Robert Hoffman, MD, Principal Investigator — Nationwide Children's Hospital; Steven T Devor, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Tjonna AE, Stolen TO, Bye A, Volden M, Slordahl SA, Odegard R, Skogvoll E, Wisloff U. Aerobic interval training reduces cardiovascular risk factors more than a multitreatment approach in overweight adolescents. Clin Sci (Lond). 2009 Feb;116(4):317-26. doi: 10.1042/CS20080249. PMID 18673303
- [Result] Tyldum GA, Schjerve IE, Tjonna AE, Kirkeby-Garstad I, Stolen TO, Richardson RS, Wisloff U. Endothelial dysfunction induced by post-prandial lipemia: complete protection afforded by high-intensity aerobic interval exercise. J Am Coll Cardiol. 2009 Jan 13;53(2):200-6. doi: 10.1016/j.jacc.2008.09.033. PMID 19130989
- [Result] Haram PM, Kemi OJ, Lee SJ, Bendheim MO, Al-Share QY, Waldum HL, Gilligan LJ, Koch LG, Britton SL, Najjar SM, Wisloff U. Aerobic interval training vs. continuous moderate exercise in the metabolic syndrome of rats artificially selected for low aerobic capacity. Cardiovasc Res. 2009 Mar 1;81(4):723-32. doi: 10.1093/cvr/cvn332. Epub 2008 Dec 1. PMID 19047339
- [Result] Ciolac EG, Bocchi EA, Bortolotto LA, Carvalho VO, Greve JM, Guimaraes GV. Effects of high-intensity aerobic interval training vs. moderate exercise on hemodynamic, metabolic and neuro-humoral abnormalities of young normotensive women at high familial risk for hypertension. Hypertens Res. 2010 Aug;33(8):836-43. doi: 10.1038/hr.2010.72. Epub 2010 May 7. PMID 20448634
- [Result] Tjonna AE, Lee SJ, Rognmo O, Stolen TO, Bye A, Haram PM, Loennechen JP, Al-Share QY, Skogvoll E, Slordahl SA, Kemi OJ, Najjar SM, Wisloff U. Aerobic interval training versus continuous moderate exercise as a treatment for the metabolic syndrome: a pilot study. Circulation. 2008 Jul 22;118(4):346-54. doi: 10.1161/CIRCULATIONAHA.108.772822. Epub 2008 Jul 7. PMID 18606913
- [Result] Moghadasi M, Mohebbi H, Rahmani-Nia F, Hassan-Nia S, Noroozi H, Pirooznia N. High-intensity endurance training improves adiponectin mRNA and plasma concentrations. Eur J Appl Physiol. 2012 Apr;112(4):1207-14. doi: 10.1007/s00421-011-2073-2. Epub 2011 Jul 17. PMID 21769734
- [Result] Giordano P, Del Vecchio GC, Cecinati V, Delvecchio M, Altomare M, De Palma F, De Mattia D, Cavallo L, Faienza MF. Metabolic, inflammatory, endothelial and haemostatic markers in a group of Italian obese children and adolescents. Eur J Pediatr. 2011 Jul;170(7):845-50. doi: 10.1007/s00431-010-1356-7. Epub 2011 Jan 6. PMID 21210148
- [Result] Hopkins ND, Stratton G, Tinken TM, McWhannell N, Ridgers ND, Graves LE, George K, Cable NT, Green DJ. Relationships between measures of fitness, physical activity, body composition and vascular function in children. Atherosclerosis. 2009 May;204(1):244-9. doi: 10.1016/j.atherosclerosis.2008.09.004. Epub 2008 Sep 9. PMID 18930229
- [Result] Kelly AS, Wetzsteon RJ, Kaiser DR, Steinberger J, Bank AJ, Dengel DR. Inflammation, insulin, and endothelial function in overweight children and adolescents: the role of exercise. J Pediatr. 2004 Dec;145(6):731-6. doi: 10.1016/j.jpeds.2004.08.004. PMID 15580192
- [Result] McMurray RG, Zaldivar F, Galassetti P, Larson J, Eliakim A, Nemet D, Cooper DM. Cellular immunity and inflammatory mediator responses to intense exercise in overweight children and adolescents. J Investig Med. 2007 Apr;55(3):120-9. doi: 10.2310/6650.2007.06031. PMID 17481381
- [Result] Meyer AA, Kundt G, Lenschow U, Schuff-Werner P, Kienast W. Improvement of early vascular changes and cardiovascular risk factors in obese children after a six-month exercise program. J Am Coll Cardiol. 2006 Nov 7;48(9):1865-70. doi: 10.1016/j.jacc.2006.07.035. Epub 2006 Oct 17. PMID 17084264
- [Result] Norris AL, Steinberger J, Steffen LM, Metzig AM, Schwarzenberg SJ, Kelly AS. Circulating oxidized LDL and inflammation in extreme pediatric obesity. Obesity (Silver Spring). 2011 Jul;19(7):1415-9. doi: 10.1038/oby.2011.21. Epub 2011 Feb 17. PMID 21331062
- [Result] Pedrosa C, Oliveira BM, Albuquerque I, Simoes-Pereira C, Vaz-de-Almeida MD, Correia F. Metabolic syndrome, adipokines and ghrelin in overweight and obese schoolchildren: results of a 1-year lifestyle intervention programme. Eur J Pediatr. 2011 Apr;170(4):483-92. doi: 10.1007/s00431-010-1316-2. Epub 2010 Oct 19. PMID 20957391
- [Result] Reinehr T, Kiess W, de Sousa G, Stoffel-Wagner B, Wunsch R. Intima media thickness in childhood obesity: relations to inflammatory marker, glucose metabolism, and blood pressure. Metabolism. 2006 Jan;55(1):113-8. doi: 10.1016/j.metabol.2005.07.016. PMID 16324929